CLINICAL TRIAL: NCT07079436
Title: Electrical Impedance Tomography (EIT) to Evaluate the Effect of Different Concentrations of Ropivacaine on Pulmonary Ventilation Function During Intercostal Nerve Blockade
Brief Title: EIT Evaluation of Pulmonary Ventilation With Different Ropivacaine Concentrations in Intercostal Nerve Blockade
Acronym: EIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jun Zhang, Doc., Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XTJLBTNDLPKA-1
Record Dates: First submitted 2025-06-03; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Intercostal Nerve Block; Pulmonary Ventilation; Anesthesia, Local; Breast Neoplasms; Surgical Procedures, Operative
Keywords: Ropivacaine; Intercostal Nerve Block; Pulmonary Ventilation Function; Electrical Impedance Tomography; Anesthetic Concentration; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: 0.25% Ropivacaine for Intercostal Nerve Blockade (Experimental): The in-plane technique was adopted, with the needle inserted 5 mm away from the long axis of the probe. During the operation, the long axis of the needle and the needle tip were displayed in real time. When the needle tip reached the extrapleural space, between the internal intercostal muscle (internal intercostal membrane) and the innermost intercostal muscle at the lower edge of the rib, and no blood was aspirated, ropivacaine (Naropin 10ml:75mg) of corresponding concentration and volume was injected into each group. Anechoic fluid was observed to spread under the internal intercostal muscle, and as the volume of the injected fluid increased, the local parietal pleura gradually descended. Inject 4 ml of 0.25% ropivacaine into each intercostal space.
  Interventions: Drug: 0.25% ropivacaine
- Arm B: 0.375% Ropivacaine for Intercostal Nerve Blockade (Experimental): The in-plane technique was adopted, with the needle inserted 5 mm away from the long axis of the probe. During the operation, the long axis of the needle and the needle tip were displayed in real time. When the needle tip reached the extrapleural space, between the internal intercostal muscle (internal intercostal membrane) and the innermost intercostal muscle at the lower edge of the rib, and no blood was aspirated, ropivacaine (Naropin 10ml:75mg) of corresponding concentration and volume was injected into each group. Anechoic fluid was observed to spread under the internal intercostal muscle, and as the volume of the injected fluid increased, the local parietal pleura gradually descended. Inject 4 ml of 0.375% ropivacaine into each intercostal space.
  Interventions: Drug: 0.375% Ropivacaine
- Arm C: 0.5% Ropivacaine for Intercostal Nerve Blockade (Experimental): The in-plane technique was adopted, with the needle inserted 5 mm away from the long axis of the probe. During the operation, the long axis of the needle and the needle tip were displayed in real time. When the needle tip reached the extrapleural space, between the internal intercostal muscle (internal intercostal membrane) and the innermost intercostal muscle at the lower edge of the rib, and no blood was aspirated, ropivacaine (Naropin 10ml:75mg) of corresponding concentration and volume was injected into each group. Anechoic fluid was observed to spread under the internal intercostal muscle, and as the volume of the injected fluid increased, the local parietal pleura gradually descended. Inject 4 ml of 0.5% ropivacaine into each intercostal space.
  Interventions: Drug: 0.5% Ropivacaine

INTERVENTIONS:
Drug: 0.25% ropivacaine — During breast quadrantectomy, intercostal nerve block is performed at the 2nd to 6th intercostal spaces along the posterior axillary line using an in-plane technique. 4ml of 0.25% ropivacaine (prepared from Naropin, 10ml:75mg) is injected into each intercostal space. Under ultrasound guidance, the needle tip is ensured to reach the space between the internal intercostal muscle (intercostal endomysium) and the innermost intercostal muscle below the rib margin. After aspiration shows no blood, the drug is injected, and anechoic fluid can be seen diffusing below the internal intercostal muscle, with the local parietal pleura gradually descending as the injected fluid volume increases.
  Other Names: Ropivacaine Hydrochloride Injection , Naropin , AstraZeneca AB, Sweden
  Arms: Arm A: 0.25% Ropivacaine for Intercostal Nerve Blockade
Drug: 0.375% Ropivacaine — During breast quadrantectomy, intercostal nerve block is performed at the 2nd to 6th intercostal spaces along the posterior axillary line using an in-plane technique. 4ml of 0.375% ropivacaine (prepared from Naropin, 10ml:75mg) is injected into each intercostal space. Under ultrasound guidance, the needle tip is ensured to reach the space between the internal intercostal muscle (intercostal endomysium) and the innermost intercostal muscle below the rib margin. After aspiration shows no blood, the drug is injected, and anechoic fluid can be seen diffusing below the internal intercostal muscle, with the local parietal pleura gradually descending as the injected fluid volume increases.
  Other Names: Ropivacaine Hydrochloride Injection , Naropin , AstraZeneca AB, Sweden
  Arms: Arm B: 0.375% Ropivacaine for Intercostal Nerve Blockade
Drug: 0.5% Ropivacaine — During breast quadrantectomy, intercostal nerve block is performed at the 2nd to 6th intercostal spaces along the posterior axillary line using an in-plane technique. 4ml of 0.5% ropivacaine (prepared from Naropin, 10ml:75mg) is injected into each intercostal space. Under ultrasound guidance, the needle tip is ensured to reach the space between the internal intercostal muscle (intercostal endomysium) and the innermost intercostal muscle below the rib margin. After aspiration shows no blood, the drug is injected, and anechoic fluid can be seen diffusing below the internal intercostal muscle, with the local parietal pleura gradually descending as the injected fluid volume increases.
  Other Names: Ropivacaine Hydrochloride Injection , Naropin , AstraZeneca AB, Sweden
  Arms: Arm C: 0.5% Ropivacaine for Intercostal Nerve Blockade

SUMMARY:
This study aims to find out how different strengths of the anesthetic drug ropivacaine affect lung breathing function when used in intercostal nerve block (a type of local anesthesia) for breast quadrantectomy surgery. Researchers will use a non-invasive imaging technique called electrical impedance tomography (EIT) to monitor lung ventilation in real time.

Why is this study being done? Intercostal nerve block is a common anesthesia method for breast surgeries, but the ideal strength of ropivacaine that balances effective pain relief with safety for lung function is not fully clear. EIT can help measure how each drug strength affects breathing by showing changes in lung airflow.

What will happen in the study? Participants: 72 adults scheduled for breast quadrantectomy, aged 18-80, will be randomly assigned to receive one of three ropivacaine strengths (0.25%, 0.375%, or 0.5%) during intercostal nerve block.

Procedures: After anesthesia, EIT will monitor lung ventilation before and after the block. Researchers will measure:

How much each lung side contributes to breathing during quiet and deep breaths. How quickly the anesthesia works, pain levels during surgery, and any side effects (like difficulty breathing or allergic reactions).

Who can join? Adults having elective breast quadrantectomy. ASA physical status I-II (generally healthy to mildly ill). BMI <35 kg/m². No history of nerve block allergies, breathing problems, or certain lung diseases.

What are the possible benefits? The study may help doctors choose the best ropivacaine strength to ensure good pain control while minimizing risks to lung function, especially for same-day surgery patients.

What are the risks? Potential risks include rare side effects from the anesthetic (like allergic reactions or low blood pressure) or temporary breathing changes, which will be closely monitored.

How is the study designed? This is a double-blind, randomized trial (neither patients nor doctors know which drug strength is used) at Fudan University Shanghai Cancer Center.

DETAILED DESCRIPTION:
The purpose of this study is to explore the impact of different concentrations of ropivacaine on pulmonary ventilation function and anesthetic efficacy during intercostal nerve block, so as to provide a reference for clinical medication selection.

This is a single-center, prospective, randomized controlled trial, with the research subjects being patients scheduled to undergo breast quadrant resection under intercostal nerve block anesthesia. Eligible patients will be randomly assigned to three groups, receiving 0.25%, 0.375%, or 0.5% ropivacaine for intercostal nerve block respectively (4ml injected into each intercostal space, blocking the 2nd to 6th intercostal nerves). The procedure will be performed by experienced anesthesiologists under ultrasound guidance, with a double-blind design where neither the anesthesiologists nor the patients are aware of the grouping and drug concentration information.

In the study, Electrical Impedance Tomography (EIT) will be used for real-time, non-invasive monitoring of changes in patients' pulmonary ventilation function before and after the block. Meanwhile, indicators related to anesthetic efficacy such as the onset time of anesthesia and block success rate will be evaluated. The entire research process includes preoperative screening, intraoperative intervention, and postoperative follow-up, aiming to clarify the relationship between ropivacaine concentration, its impact on pulmonary ventilation function, and anesthetic efficacy, so as to provide a basis for optimizing the clinical application of ropivacaine in intercostal nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective breast quadrantectomy;
* Aged 18-80 years;
* American Society of Anesthesiologists (ASA) physical status I-II;
* Body mass index (BMI) <35 kg/m².

Exclusion Criteria:

* Contraindications for nerve block: infection at the puncture site, local anesthetic allergy, coagulation dysfunction or bleeding risk;
* Patients with unilateral diaphragmatic paralysis;
* Patients with severe ventilatory or gas exchange dysfunction;
* Complicated with acute or chronic pulmonary and bronchial diseases, sleep apnea syndrome;
* Mental disorders;
* Patients who refuse to participate;
* Patients whom the researchers consider unsuitable for the clinical trial, with reasons to be specified.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage decrease (/L) of the surgical side lung ventilation to total lung ventilation after blockade | 15 minutes after blockade
  The patient was placed in a supine position, and an EIT electrode strip was placed along the 4th intercostal space on the chest. Continuous monitoring of EIT (Drager Infinity C500, Germany) was performed, and tidal resistance changes during quiet breathing and deep breathing over at least 5 consecutive respiratory cycles were collected to construct lung ventilation distribution images. The main focus is to compare the changes in ROI% in different regions before and after the block, with comparisons made in 4 quadrants: "left upper, right upper, left lower, right lower".

SECONDARY OUTCOMES:
Block success rate | 5 minutes after surgery
  The patient was able to undergo the surgery successfully without the need for additional rescue anesthesia measures.

OTHER OUTCOMES:
Adverse events | 1 hour after surgery
  The number of cases with adverse events, adverse reactions, and serious adverse events (to be specified) such as local anesthetic toxicity, Horner's syndrome, and pneumothorax.
Pain-related assessment | 24 hours after surgery
  The Numerical Rating Scale (NRS) was used to assess the patient's pain score via telephone.
Pain-related assessment | 6 hours after surgery
  The Numerical Rating Scale (NRS) was used to assess the patient's pain score via telephone.

IPD SHARING:
Plan to Share IPD: No
Sharing is not permitted under local laws.